CLINICAL TRIAL: NCT05677035
Title: A Single-center, Open-label, Parallel-group, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LINO-1713 in Healthy Korean Female Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LINO-1713 in Healthy Korean Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT-014-01
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacokinetic evaluation (Experimental): LINO-1713 (Estetrol 15mg/Drospirenone 3mg)
  Interventions: Drug: LINO-1713 1 tablet
- Pharmacodynamic evaluation (Experimental): LINO-1713 (Estetrol 15mg/Drospirenone 3mg)
  Interventions: Drug: LINO-1713 once a day for 24 days

INTERVENTIONS:
Drug: LINO-1713 1 tablet — LINO-1713 1 tablet is administered once. Oral administration with 200mL of water
  Arms: Pharmacokinetic evaluation
Drug: LINO-1713 once a day for 24 days — Oral administration is performed with 200 mL of water. Instruct subjects to take the drug at the same time as possible.
  Arms: Pharmacodynamic evaluation

SUMMARY:
A single-center, open-label, parallel-group, phase 1 study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of LINO-1713 in healthy Korean female subjects

ELIGIBILITY:
Inclusion Criteria:

* Women with a Body Mass Index (BMI) between 18kg/m2 ~ 28kg/m2

Exclusion Criteria:

* Clinically significant cardiovascular disease, respiratory disease

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters: Cmax | Before and after administration 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144, and 168 hours
Pharmacokinetics parameters: Tmax | Before and after administration 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48, 72, 96, 120, 144, and 168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea